CLINICAL TRIAL: NCT06505213
Title: Multimodal Brain Monitoring as an Early Warning and Prognostic Tool for Acute Brain Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024070747
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Acute Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The primary aim of this study is to evaluate the effectiveness of multimodal brain monitoring technologies as both an early warning system and a prognostic tool in patients suffering from acute brain injuries. This research seeks to determine how effectively these tools can predict clinical outcomes and prevent complications by providing early alerts to healthcare professionals.

DETAILED DESCRIPTION:
Acute brain injury, including traumatic brain injury (TBI) and stroke, presents significant challenges in clinical management, primarily due to the complexity of the brain's response to injury and the critical timing required for effective intervention. Multimodal brain monitoring, which integrates various physiological data points like brain electrical activity, cerebral blood flow, and brain tissue oxygenation, offers a comprehensive view of a patient's cerebral status. This study builds on the premise that a better understanding and real-time monitoring of these variables can significantly improve patient outcomes by enabling timely and targeted interventions.

ELIGIBILITY:
Inclusion Criteria

1. Must be 18 years of age or older.
2. Diagnosed with Traumatic Brain Injury (TBI) or has suffered from acute brain injury due to intracranial hemorrhage or subarachnoid hemorrhage.
3. Defined as an admission Glasgow Coma Scale (GCS) Eye Response score of 1 (unable to open eyes) and a GCS Motor Response score of ≤5 (unable to obey commands).
4. Occurs within 48 hours of admission, where the patient does not open eyes and motor score drops to 5 or below.

Exclusion Criteria

1. Patients who were not admitted to the Intensive Care Unit (ICU) are excluded.
2. Patients with forms of acute brain injury other than those specified (TBI, intracranial hemorrhage, subarachnoid hemorrhage) are also excluded.
3. Patients with known severe liver or kidney dysfunction are excluded.
4. Patients whose vital signs are extremely unstable after admission, with a very poor prognosis and considered unable to survive, and whose family has decided to forgo further treatment.
5. Patients who had a Modified Rankin Scale greater than 2 before the onset of the current illness.
6. Patients with a history of congenital or acquired hemorrhagic diseases, coagulation factor deficiencies, or thrombocytopenic disorders.
7. Pregnant or lactating women, as well as those planning to become pregnant within the next 90 days.
8. Patients with severe psychiatric disorders or dementia who are unable to provide informed consent or complete follow-up requirements.
9. Patients who have participated in other interventional clinical trials within 30 days prior to randomization, or who are currently participating in other clinical research.
10. Any other reasons that the researcher deems unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically Ill, Acute Brain Injury Adult Patients.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Relation between multimodal brain monitoring parameters and outcome. | 6 months
  Association between advanced multimodal brain monitoring parameters of the first 48h of admission and six months functional outcome (Glasgow Outcome Score Extended)

SECONDARY OUTCOMES:
Neuromonitoring Pattern | 3-5 days
  Describe multimodal neuromonitoring parameters variation and identify trends.
Neuromonitoring and Short Term Outcome | 28 days
  Association between advanced multimodal brain monitoring parameters and 28 days functional outcome (Glasgow Outcome Score Extended)